CLINICAL TRIAL: NCT06096532
Title: Adipose Tissue Blood Flow in Aging Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kelli A. Lytle, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-004200; UL1TR002377 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older Adults (Other)
  Interventions: Other: 75 gm oral glucose load
- Younger Adults (Active Comparator)
  Interventions: Other: 75 gm oral glucose load

INTERVENTIONS:
Other: 75 gm oral glucose load — Consumption of 75 gm oral glucose load in order to test nutrient responsiveness

SUMMARY:
The goal of this basic science clinical trial is to understand whether adipose tissue blood flow changes between younger and older healthy adults.

The main question[s] it aims to answer are:

* Is basal and nutrient responsive adipose tissue blood flow (ATBF) different between younger and older adults
* What molecular and systemic signatures related to adipose tissue blood flow are altered between these two groups.

Participants will undergo measurements of adipose tissue blood flow using the xenon washout technique, undergo 2 abdominal subcutaneous adipose tissue biopsies, and drink a sugary drink.

DETAILED DESCRIPTION:
On Visit 1, volunteers will provide written informed consent (and urine pregnancy test for women of childbearing age), complete a Dual x-ray absorptiometry scan, baseline labs (comprehensive metabolic panel) and a cardiopulmonary exercise test. Participants will arrive fasted at 08:00, and urine pregnancy test for women of childbearing age administered and an intravenous catheter will be placed. Following 30min of supine rest, baseline venous blood samples will be collected. ATBF will be assessed on participants' left abdomen first by measurement of blood flow using 133Xenon washout method. Immediately thereafter, an abdominal adipose tissue biopsy of the left side will be performed but ≥6 cm distant from location of 133Xenon injections. Subjects will them consume 75 gm glucose; because ATBF peaks 30-60 minutes following ingestion of glucose, ATBF measures will start 30 minutes after ingestion on the contralateral side followed immediately by plasma measures and another adipose tissue biopsy. During ATBF measurements, brachial blood pressure will be assessed in two-minute intervals.

ELIGIBILITY:
Inclusion criteria

* Within the ages of 18-35 years or 65-80 years at time of study visit
* BMI between 20-25.0 kg/m2.

Exclusion criteria:

* Presence of diagnosed cardiometabolic diseases (e.g., Type 2 diabetes, hypertension, Heart Failure)
* Taking prescription anticoagulants
* Taking prescriptions or supplements that effect adipose tissue metabolism (i.e., statins, Thiazolidinediones, niacin, atypical antipsychotics, or fish oil)
* Pregnant or nursing
* Inability to provide written informed consent
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue blood flow | Baseline, pre-intervention fasting and immediately following 75 gm oral glucose load
  blood flow will be measured in the upper body subcutaneous adipose tissue using 133 Xenon washout and reported as blood flow in ml/min/100g adipose tissue.

SECONDARY OUTCOMES:
Genomic alterations | Baseline, pre-intervention fasting and immediately following 75 gm oral glucose load
  RNA-Seq from adipose tissue biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Lytle, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials